CLINICAL TRIAL: NCT07044141
Title: Efficacy of Oral Tofacitinib in Combination With Narrow Band UVB in the Treatment of Vitiligo
Brief Title: Efficacy of Oral Tofacitinib in Combination of Narrow Band UVB in Treatment of Vitiligo
Acronym: NB-UVB
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Dr ayesha wahid, Dr saadiya siddiqui, Lahore General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dermatology LGH
Record Dates: First submitted 2025-06-23; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-05

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Azathioprine; tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Azathioprine is an immunomodulator used in treatment of vitiligo
  Interventions: Drug: Azathioprine
- Group B (Active Comparator): Tofacitinib It is a Janu kinase pathway inhibitor
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Azathioprine — azathioprine 50mg twice daily will be given
  Arms: Group A
Drug: Tofacitinib — It is a janus kinase inhibitor
  Arms: Group B

SUMMARY:
20 patients will be enrolled. All were given narrowband UVB . 10 wil be give oral azathriopfine . 10 will be given tofacitinib

DETAILED DESCRIPTION:
Total 20 patients will be enrolled. All were given narrowband UVB . 10 wil be give oral azathriopfine 50mg twice daily. 10 will be given tofacitinib 5mg twice daily. For 6 months

ELIGIBILITY:
Inclusion Criteria:

* patient of vitiligo with any VASI both genders 18 to 60yrs

Exclusion Criteria:

* pregnancy/lactation Hyerlipidrmia Patient on immunemodulator Histry pf tuberculosis Immunocompromised patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
VASI improvement upto 50% | 6 months
  Study will be considered efficacious if 50% improvement in VASI from baseline is seen by end of 6 months of study

CONTACTS AND LOCATIONS:
Locations (1):
- Lahore general.hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided